CLINICAL TRIAL: NCT03559972
Title: Open-Label, Randomized, Multi-center Study to Evaluate the Efficacy and Tolerability of Two Topical Regimens in Subjects With Moderate to Severe Facial Photodamage Who Have Received Cosmetic Injections
Brief Title: Study to Evaluate Efficacy and Tolerability of Two Topical Regimens in Subjects With Moderate to Severe Facial Photodamage Who Have Received Cosmetic Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKM18-HULK-INJ
Record Dates: First submitted 2018-05-23; First posted 2018-06-18 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Facial Photodamage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group #1 (Experimental): Subject in Treatment group 1 will apply the following products in the morning and evening.
  1. SkinMedica Facial Cleanser
  2. Hulk (cosmetic investigational)
  3. Marvel AM (cosmetic investigational)
  4. Marvel PM (cosmetic investigational)
  5. SkinMedica HA5 Rejuvenating Hydrator
  6. SkinMedica Rejuvenative Moisturizer
  7. SkinMedica Essential Defense Mineral Shield SPF 35 Sunscreen
  Interventions: Other: on-label facial injection
- Treatment group #2 (Experimental): Subject in Treatment group 2 will apply the following products in the morning and evening.
  1. SkinMedica Facial Cleanser
  2. SkinMedica TNS Essential Serum
  3. Marvel AM (cosmetic investigational)
  4. Marvel PM (cosmetic investigational)
  5. SkinMedica HA5 Rejuvenating Hydrator
  6. SkinMedica Rejuvenative Moisturizer
  7. SkinMedica Essential Defense Mineral Shield SPF 35 Sunscreen
  Interventions: Other: on-label facial injection

INTERVENTIONS:
Other: on-label facial injection — Assessing if adding SkinMedica's cosmetic topical skincare regimens improves the appearance of the skin and the subject's experience, when used after pre-elected on-label facial injection

SUMMARY:
This study will assess the efficacy and tolerability of two topical regimens (containing cosmetic human fibroblast-derived, physiologically-balanced growth factor combination products (HULK and TNS Essential Serum)

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 30 years and older with Fitzpatrick skin type I-VI
* Pre-elected to receive on-label facial injection(s) (i.e. neuromodulator injection and/or filler injections)
* Experienced injection patients defined as having received at least 1 facial injection in the past 2 years.
* Current users of non-physician-dispensed brand skin care products (i.e. only using products that are available at drugstores or department stores
* Good general health and free of any disease state or physical condition (e.g. psoriasis, rosacea, scars, tattoos etc.)
* Willingness to have exams and digital photos performed on the face.
* Willingness to cooperate and participate by following study requirements (including using the provided test products) for the duration of the study and to report any adverse event symptoms or reactions immediately.
* Willingness to discontinue use of their current skincare products starting at their Week 4 visit in this study.
* Willingness to not use any other products, including self-tanners, on their face for the duration of the study other than make-up with an established tolerance of at least 1 month.
* Willingness to withhold all facial treatments during the course of the study including microdermabrasion, peels, facials, laser treatments and tightening treatments.
* .Willingness to avoid as much as possible, direct and prolonged sun exposure for the duration of the study (including tanning beds), especially from 10 AM to 2 PM. Subjects are asked to wear protective clothing prior to and during exposure.
* If of child-bearing potential, willing to use an acceptable method of contraception throughout the study. Acceptable methods of birth

Exclusion Criteria:

* Who are nursing, pregnant, or planning to become pregnant during the study according to subject self-report.
* Individuals with active symptoms of allergy, cold sore or warts, active psoriasis or eczema, rosacea, sunburn, open wounds, neurotic excoriations, excessive scarring, tattoos, or other skin conditions in the test areas that would interfere with the assessments of this study.
* Uncontrolled disease such as diabetes, hypertension, hyper or hypo-thyroidism, active hepatitis, immune deficiency, or autoimmune.
* Individuals who have a pre-existing or dormant dermatologic condition (e.g., psoriasis, atopic dermatitis, rosacea, skin cancer, etc.)
* Individuals who require electrolysis, waxing, or use depilatories on the face during conduct of the study.
* Individuals with any planned surgeries and/or invasive medical procedures during the course of the study
* Individuals who are currently participating in any other facial usage study or have participated in any clinical trial within 4 weeks prior to inclusion of the study.
* Subjects currently on or planning to participate on any type of research study at another facility or a doctor's office during this study.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Clinical grading of the full face on the Griffith's modified 10-point scale | Baseline, Week 4, Week 16
  Investigator will assess the following parameters on a Griffith's modified 10-point scale (0 = None, 1 to 3 = Mild, 4 to 6 = Moderate, 7 to 9 = Severe)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Makino, Study Director — Allergan
Locations (2):
- United States (2):
  - Cosmetic Laser Dermatology, San Diego, California
  - Suzanne Bruce and Associates, PA, The Center for Skin Research, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance — http://www.allerganclinicaltrials.com/